CLINICAL TRIAL: NCT00385021
Title: ChronoFOLFOX Plus Avastin for Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Southwestern Regional Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTCT 06-06
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Colorectal Neoplasms
Keywords: Advanced; metastatic; colorectal; cancer; Avastin
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 5-Fluorouracil, leucovorin, oxaliplatin, avastin

SUMMARY:
To determine efficacy in the delivery of chronomodulated chemotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to determine if treatment with 5-Fluorouracil, leucovorin, oxaliplatin, and Avastin will cause colorectal tumor cells to shrink or disappear. The study will also determine the safety of these drugs when given together and the quality of life of the patients who are enrolled in the study.

It is thought that these drugs will be better tolerated if they are chronomodulated, i.e., if they are given at certain times of day rather than as a continuous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of adenocarcinoma in primary colon or rectum tumor.
* Evidence of metastatic colorectal cancer or loco-regional recurrence or unresectable disease.
* Ages 18 to 86 years.
* Presence of at least one bi-dimensionally measurable disease with at least one diameter > or = 2 cm.
* WHO/ECOG performance status < 3 (0, 1, or 2)
* Prior treatment with oxaliplatin, 5-FU, or leucovorin permitted.
* Signed informed consent

Exclusion Criteria:

* Peripheral sensory neuropathy > or = grade 3.
* Serum bilirubin (total) > 3 X ULN.
* Symptomatic or uncontrolled brain metastasis.
* Metastases limited to bone, pleural effusion, or ascites.
* Uncontrolled overt cardiac disease.
* Uncontrolled hypercalcemia.
* Uncontrolled infections.
* Uncontrolled hypertension (>180/110)
* History of GI perforation.
* History of arterial thromboembolic events.
* History of congestive heart failure.
* Patients taking warfarin (Coumadin).
* Patients who are pregnant.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine if the rate of adverse events among patients receiving chronoFOLFOX plus Avastin is acceptable compared to that in previous studies using the FOLFOX4 regimen. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Petra Ketterl, MD, Principal Investigator — Cancer Treatment Centers of America at Southwestern Regional Medical Center, Inc.
Locations (1):
- Cancer Treatment Centers of America at Southwestern Regional Medical Center, Inc., Tulsa, Oklahoma, United States